CLINICAL TRIAL: NCT04531488
Title: Powered Mobility Training of Children With Special Needs: Conventional Versus Simulator-based Practice
Brief Title: Simulator Based Powered Mobility Training of Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Naomi Gefen, Naomi Gefen, Deputy Director General, Principal Investigator, Alyn Pediatric & Adolescent Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004-17
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Cerebral Palsy
Keywords: Powered mobility; Simulator; Powered Mobility Outcome Measures
MeSH Terms: conditions — Cerebral Palsy | interventions — Wheelchairs

STUDY DESIGN:
Intervention Model Description: Two groups that practiced powered mobility via different modes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powered Mobility Training Simulator (Experimental): Powered mobility simulator- the McGill Immersive Wheelchair Simulator (MiWe) was developed for adults. In a previous study the simulator was found valid for use with children. Participants were provided a laptop, joystick and the software program- MiWe- to practice at home or school
  Interventions: Procedure: Powered Mobility Training Simulator
- Training with Powered Wheel Chair (Active Comparator): Participants were provided with a powered wheelchair to practice at home or school
  Interventions: Other: Training with Powered Wheel Chair

INTERVENTIONS:
Procedure: Powered Mobility Training Simulator — Two groups of participants- 18 in each- were provided with either a simulator or powered wheelchair. Both groups were tested at baseline for powered mobility level. Both groups the practiced at home or school for 12 weeks, 4 times a week for at least 20 minutes. Both groups returned and underwent another evaluation to assess powered mobility level after 12 weeks of practice.
  Other Names: Powered Mobility Training with Wheel Chair
  Arms: Powered Mobility Training Simulator
Other: Training with Powered Wheel Chair — Training with Powered Wheel Chair
  Arms: Training with Powered Wheel Chair

SUMMARY:
This study compared conventional powered mobility practice to simulator based practice of children with special needs aged 6-18 years.

DETAILED DESCRIPTION:
This study compared conventional powered mobility practice to simulator based practice of children with special needs aged 6-18 years.

The study has 3 stages: 1) Simulator validity study 2) Powered mobility outcome measures reliability and validity for children 6-18 years 3) Intervention study to compare simulator based practice and powered mobility practice.

1. Simulator validity study included 30 children aged 6-18 years, proficient powered mobility drivers. All participants had physical disabilities- CP or Neuromuscular conditions.
2. This stage included the first 30 children from the intervention study. Data for the study was based on the first evaluation out of the two evaluations in the study.
3. This stage included 36 children aged 6-18 years in need of powered mobility practice to become a proficient driver. The particpants were divided into two groups- experimental (simulator based practice) and control group (standard powered wheelchair practice).

ELIGIBILITY:
Inclusion Criteria:

* Children with a physical disability that are not proficient powered mobility driver
* Children that can use a joystick

Exclusion Criteria:

* Children with visual accuracy limitations that cannot be corrected with glasses or contact lens;
* Children who have a severe intellectual and developmental disability as defined by the Israel Ministry of Welfare's index for intellectual and developmental disabilities and reported by parents; Children that have a unstable medical conditions that prevent them from participating in powered mobility training (e.g., epilepsy)
* Children that can operate a powered wheelchair via switches or a scanning device.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Powered Mobility Program- Assessing change from Baseline to End of intervention | This outcome measure is done at baseline and after 12 weeks of practice.
  This is an evaluation that has up to 34 items that assess the driving skills of powered wheelchair users. Each skill can receive a score of 0-5. The higher the score the better. The total sum of all skills is divided by the number of skills tested and an average score ranging from 0-5 is recorded.
Assessment of Learning Powered Mobility Use- Assessing change from Baseline to End of intervention | This outcome measure is done at baseline and after 12 weeks of practice.
  This is an evaluation that has 8 levels of 5 skills. It assess the level of powered mobility driving in areas that the PMP does not- cognitive, emotional, social. Each of the 5 skills receives a score of 1-8. The sum of all skills scores is divided by 5. The score can be between 1-8. A higher score is better.
The Israel Ministry of Health Proficiency Test- Assessing change from Baseline to End of intervention | This outcome measure is done at baseline and after 12 weeks of practice.
  This is an evaluation that assess 7 powered mobility skills. The driver needs to succeed 4/5 times each skill in order to pass test. Each of the 7 skills receives a score of 1,3,5. The sum of all skills is divided by 7 and the average score is recorded 1-5. The higher the score the better.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Gefen, M.A., Principal Investigator — Alyn Pediatric and Adolescent Rehabilitation Hospital
Locations (1):
- Alyn Pediatrics Rehabilitation Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Gefen N, Archambault PS, Rigbi A, Weiss PL. Pediatric powered mobility training: powered wheelchair versus simulator-based practice. Assist Technol. 2023 Sep 3;35(5):389-398. doi: 10.1080/10400435.2022.2084183. Epub 2022 Jun 23. PMID 35737961